CLINICAL TRIAL: NCT03553381
Title: Oxidative Stress, Inflammation, and Lipoprotein Chemical Composition in Obesity and Metabolic Syndrome: Effects of Diet-induced Weigh Loss
Brief Title: Oxidative Stress, Inflammation, and Lipoprotein in Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: roberta cazzola (Other)
Collaborators: Luigi Sacco University Hospital (Other); Istituti Clinici di Perfezionamento di Milano (Other)
Responsible Party: Sponsor-Investigator, roberta cazzola, Principal Investigator, University of Milan
Organization: University of Milan (Other)
Other Study IDs: RV_RIC_AT16RCAZZ
Record Dates: First submitted 2018-05-22; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Metabolic Syndrome; Obesity, Metabolically Benign
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Metabolically Benign

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasma and serum, and erythrocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese without MS: BMI 25- 35 Kg/mq without metabolic syndrome (MS) submitted to hypocaloric balanced diet
  Interventions: Other: hypocaloric balanced diet
- obese with MS: BMI 25- 35 Kg/mq with metabolic syndrome submitted to hypocaloric balanced diet
  Interventions: Other: hypocaloric balanced diet

INTERVENTIONS:
Other: hypocaloric balanced diet

SUMMARY:
Obesity is associated with general low grade inflammation and, consequently, of oxidative stress that affects properties and functionality of lipoproteins. Metabolic syndrome exacerbate low grade inflammation. The intentional weight loss of at least 5% of the initial weight can modulate the pro-inflammatory state and reduce the oxidative stress related to the metabolic syndrome, thus diminishing the cardiovascular risk.

DETAILED DESCRIPTION:
Metabolic syndrome is a clustering of risk factors for the development of cardiovascular disease and type 2 diabetes mellitus. Patients with metabolic syndrome have an increased general low grade inflammation and, consequently, of oxidative stress that affects properties and functions of lipoproteins (Dandona et al 2005). Intentional weight loss can improve or prevent many of the metabolic syndrome-related risk factors and these benefits are often found after weight loss of at least 5% of initial weigh.

Aim: i) to investigate the structure and functionality of plasma lipoproteins, oxidative stress and the inflammatory condition in subjects with BMI between 25kg/mq and 35 kg/mq and with or without metabolic syndrome; and ii) to test the effects of weight loss of at least 5% of initial weigh promoted by an hypo-caloric balanced diet on these parameters.

Methods: Eighty overweight and moderately obese subjects (BMI: 25 - 35 kg/m2) with or without metabolic syndrome were recruited for the study. Fasting blood samples were taken and analyzed for routine laboratory analysis, lipoprotein isolation and analysis, and oxidative stress and inflammation markers measurements. The subjects received an hypo-caloric balanced diet. Fasting blood samples were taken from subjects who had lost at least 5% of their initial weight at the end of the intervention period and analyzed for same markers determined at baseline.

ELIGIBILITY:
1. Inclusion Criteria.

1.a Group "Obese with MS":

* BMI between 25 e 35 Kg/m2
* presence at least three of the following:1) waist circumference >102 cm for males or > 88 cm for females; 2) triglycerides: ≥ 150 mg/dL;3) HDL-cholesterol < 40 mg/dL in males or < 50 mg/dL in females; 4) hypertension (systolic blood pressure ≥ 130 mm Hg or diastolic blood pressure ≥ 85 mm Hg or antihypertensive intake); 5) glycemia: ≥ 110 mg/dL
* Alcohol consumption < 25 g/die
* No smoking or smoking less that 5 cigarettes/die
* No use of antioxidant based supplements
* Absence of hormonal treatments
* Informed consent signature

  1.b Group "Obese without MS":
* BMI between 25 e 35 Kg/m2
* Alcohol consumption < 25 g/die
* No smoking or smoking less that 5 cigarettes/die
* No use of antioxidant based supplements
* Absence of hormonal treatments
* Informed consent signature

  2. Exclusion Criteria
* Presence of major disease
* Receiving hypoglycemic treatment
* Receiving treatments that alter lipoprotein metabolism
* Receiving hormonal treatments
* Use of antioxidant supplement
* Alcohol consumption > 25 g/die
* Smoking > 5 cigarettes/die.
* For women:pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects were males and females overweight or moderately obese with or without metabolic syndrome on a calorie-controlled diet.
  Those that lost at least 5% of the initial weight were analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-12-30 (Actual); Primary Completion 2012-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Lipoprotein and plasma oxidizability | six months
  kinetics of 2,2'-diazobis-(2-amidinopropane)-dihydrochloride (AAPH)- induced peroxidation of plasma, LDL or HDL labeled with fluorescent probes. The length of the lag phase (lag-time) and the velocity of the reaction in the propagation phase (slope) of peroxidation kinetic curves are used as indices of sample oxidizability
Oxygen Reactive Species (ROS) | six months
  plasma levels of ROS (mg/dL)
Inflammatory markers | six months
  Plasma levels of cytokines (pg/ml);

SECONDARY OUTCOMES:
Lipoprotein chemical composition | six months
  Levels of proteins (mg/dL), triacylglycerol (mg/dL), free and esterified cholesterol (mg/dL) and phospholipids (mg/dL) of very low density lipoprotein (VLDL), LDL and HDL.
Cholesteryl ester transfer protein (CETP) | six months
  Plasma levels of CETP (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Cazzola, PhD, Principal Investigator — University of Milan
Locations (2):
- Italy (2):
  - ASST Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO, Milan
  - Ospedale "L. Sacco" - ASST Fatebenefratelli Sacco, Milan

REFERENCES:
- [Background] Dandona P, Aljada A, Chaudhuri A, Mohanty P, Garg R. Metabolic syndrome: a comprehensive perspective based on interactions between obesity, diabetes, and inflammation. Circulation. 2005 Mar 22;111(11):1448-54. doi: 10.1161/01.CIR.0000158483.13093.9D. No abstract available. PMID 15781756